CLINICAL TRIAL: NCT00587795
Title: Orthopedic Study of the Aircast StabilAir Wrist Fracture Brace
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to enroll subjects
Sponsor: Mayo Clinic (Other)
Collaborators: AirCast LLC (Industry)
Responsible Party: Principal Investigator, David Dennison, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 228-06
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-04

CONDITIONS: Radius Fractures
MeSH Terms: conditions — Radius Fractures | interventions — Casts, Surgical

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- StabilAir Wrist Brace (Active Comparator): One study group will consist of patients treated with the StabilAir Wrist Brace.
  Interventions: Device: StabilAir Wrist Brace
- Control (Placebo Comparator): Study arm will consist of patients that are treated with placement of sugar tong splint or plaster cast.
  Interventions: Other: Placement of sugar tong splint or plaster cast

INTERVENTIONS:
Device: StabilAir Wrist Brace — Patient will be placed in a StabilAir Wrist Brace 10-14 days after initial injury and return for follow up visits at 6 weeks; 3, 6, 12 and 24 months.
  Arms: StabilAir Wrist Brace
Other: Placement of sugar tong splint or plaster cast — Patients will receive a sugar tong splint or plaster cast for their wrist fracture. They will return for x-rays and an exam at 6 weeks; 3, 6, 12 and 24 months.
  Other Names: Sugar tong splint or plaster cast
  Arms: Control

SUMMARY:
Objectives:

- To obtain clinical evidence for the safety and efficacy in using the StabilAir Wrist Fracture Brace for the following cases:

1. Acute (emergency department) treatment of non-displaced, stable extra- articular distal radius fractures;
2. To obtain comparative data between traditional therapies (sugar tong, plaster backslab, long arm or short arm cast) and the use of the StabilAir brace for each patient qualified by specific criteria.

Hypothesis:

1) For stable, non-displaced fractures, the StabilAir Brace is as effective as a sugar tong splint in the acute setting. 2) In cases where full forearm immobilization is initially preferred, the StabilAir is effective as a follow-up to sugar tong splitting once the need for full immobilization has passed.

DETAILED DESCRIPTION:
Data Collection and Study Design:

This will be a single center, prospective, randomized controlled trial. The investigators planned to collect data from 80 patients with undisplaced distal radius fractures. Half were to be treated with the plastic back slab or sugar tong splint (if there were an ulnar styloid fracture) and half were to be treated with the StabilAir splint. The initial treatment, which was to occur upon the patient's arrival at the emergency room and prior to study randomization, required full forearm and wrist immobilization in the acute phase treated with sugar tong splinting. At the patient's follow-up visit, which was to happen ≤10 days post injury and initial evaluation, when it was determined that full forearm immobilization was no longer necessary, patients were informed of the study, consented, and randomized (as in the flip of a coin) to one of the two study groups using a computerized randomization process that was controlled by the study coordinator. One study group was to consist of patients treated with either sugar tong splint or plaster casting and the other study group was to consist of patients treated with the StabilAir brace. Throughout entire study, the sugar tong splint/casting patients was to be the control group.

Patients were to be asked to return for the following visits after they were randomized:

* 10-14 days post randomization
* 35 to 42 days (5 to 6 weeks) post randomization
* 77 to 84 days (11 to 12 weeks) post randomization;
* And at 12 and 24 months.

At each visit they were to have x-rays of their wrist and an exam with the physician. In addition, they were to be asked to complete questionnaires regarding their general health, daily activities and pain.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females Age ≥ 18 yrs
* Undisplaced distal radial fractures (with/without ulnar styloid fractures)

Exclusion Criteria:

* Age < 18 yrs
* Intra-articular fracture - displaced
* Loss of reduction after cast or brace treatment
* Excessive comminution (> 50% metophysis)
* Failed closed reduction (CR) (Unacceptable alignment status post CR: Short >2mm; Dorsal angulation >0° (neutral), Radial inclination < 15°)
* Ipsilateral ulna fractures (not styloid)
* Open fracture
* Senile or dementia or lack of understanding of treatment
* Previous fracture distal radius
* Patients with displaced fractures that require pin fixation, external fixation, plate fixation or who qualify for "crystalline injection fracture healing protocol" are excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-04; Primary Completion 2008-08 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G Dennison, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One subject was recruited from the Mayo Clinic in Rochester, Minnesota in 2007.
Period: Overall Study
Arm/Group | StabilAir Wrist Brace | Control
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | StabilAir Wrist Brace | Control | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Distal Radius Fracture at 8 Weeks
Description: The investigators planned to make radiographic assessments using the Stewart Score. The Stewart Score can range from 1 to 12, with a higher score indicating poor function: excellent (0), good (1-3), fair (4-6) and poor (7-12).
Time Frame: baseline, 8 weeks
Arm/Group | StabilAir Wrist Brace | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | StabilAir Wrist Brace | Control
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
Early termination due to inability to enroll subjects, and concern about subject compliance in the use of the Stabilair wrist brace. The one subject enrolled disliked the brace and quickly withdrew from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes